CLINICAL TRIAL: NCT02631356
Title: The Effect of Succinylated Gelatin on the Blood Viscosity and Oxygen Delivery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Feng Xia, Professor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2015[22]
Record Dates: First submitted 2015-11-24; First posted 2015-12-16 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Blood Viscosity
MeSH Terms: interventions — Ringer's Lactate; succinylated gelatin

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Ringer's lactate solution (Placebo Comparator): Infusion of Ringer's lactate solution (10ml/kg) in the control group
  Interventions: Drug: Ringer's lactate solution
- Succinylated gelatin (Active Comparator): Infusion of Succinylated gelatin (10ml/kg) in the test group
  Interventions: Drug: Succinylated gelatin

INTERVENTIONS:
Drug: Ringer's lactate solution
  Arms: Ringer's lactate solution
Drug: Succinylated gelatin
  Arms: Succinylated gelatin

SUMMARY:
The study is to investigate the effect of succinylated gelatin on the blood viscosity and oxygen delivery in patients during surgeries, so as to have a better understanding of the safety in the use of succinylated gelatin for surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 years and 60 years
* ASA physical status I and II
* surgical procedures requiring general anesthesia with continuous CVP and arterial pressure monitoring

Exclusion Criteria:

* Patients younger than 16 y or older than 60 y
* Body Mass Index (BMI) <18 or >30
* Allergy to any of the drugs used
* Severe cardiovascular dysfunction
* Patient refusal

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
The patient's arterial blood viscosity (mpa.s) as tested by viscometer | up to 5 months (after the infusion of succinylated gelatin )

SECONDARY OUTCOMES:
The patient's oxygen delivery index (DO2I) as calculated by Vigileo | up to 5 months (after the infusion of succinylated gelatin )

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China